CLINICAL TRIAL: NCT04657419
Title: Fatigue and Sleep in Patients With COVID-19
Acronym: COFATSOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/52
Record Dates: First submitted 2020-12-07; First posted 2020-12-08 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; fatigue
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant: Patient or health professional coming to the Bordeaux University Hospital screening center for COVID-19 screening
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — Self-questionnaires will be completed by the participants :
  * General health and mental health
  * Fatigue
  * Burn-Out
  * Sleepiness
  * Sleep hygiene
  * Symptoms of COVID

SUMMARY:
Recent studies show that patients who have contracted COVID-19 retain very significant fatigue after resolving the infectious episode. This fatigue may be explained by low-grade inflammation. There is more data for patients with COVID-19 who have been hospitalized than for non-hospitalized patients with milder forms.

However, COVID-19 related fatigue would not only affect elderly people with severe cardiopulmonary consequences but also young subjects without severities. This notion is not very widespread and to date, COVID contracted by young subjects is considered to have very few consequences on their health.

It is also known that the prevalence of sleep debt is significant in the general population and particularly in young people, and it is also known that sleep deprivation increases low-grade inflammation and facilitates the risk of viral contamination. The association between sleep deprivation, drowsiness and possibly low-grade inflammation raise questions about the mechanisms of fatigue in the general population.

Investigators are also entitled to wonder to what extent the chronic sleep debt suffered by the French population can explain an increased risk of contamination by COVID 19 but also significant residual fatigue after COVID infection.

Bordeaux University Hospital screens 2,000 subjects per day at risk of being infected by COVID, it would be very interesting to measure, in a population of young adults aged 18-45 years, frequently exposed to a sleep debt, sleep hygiene (bedtime and wake-up times, sleep and wake-up schedules, and overall sleep satisfaction), average sleep duration, level of fatigue and drowsiness and to compare these thresholds between subjects with or without COVID 19 according to nasopharyngeal PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patient or healthcare professional going to screening center to perform a PCR test for COVID-19
* Between 18 and 45 years old
* Symptomatic or not
* Whether or not COVID-19 contact-case
* Accepting to participate to the research
* Informed and having expressly transmitted their non-opposition to participate in the study

Exclusion Criteria:

* Participants who do not speak French or who cannot read or write
* Patients who do not have contact information for recall
* Refusal to participate in the study.
* Majors under guardianship or curatorship.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient or healthcare professional going to screening center to perform a PCR test for COVID-19
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | one month after inclusion (T0)
  Presence of significant fatigue as measured by the Fatigue Severity Scale (FSS) at 1 month.
  Score from 1 to 7 FSS is a 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree.
  The minimum score is 9 and maximum score possible is 63. Higher is the score, greater is the fatigue severity

SECONDARY OUTCOMES:
COVID Diagnosis | inclusion (T0)
  Diagnosis of COVID-19 by nasopharyngeal PCR
Fatigue evolution | Inclusion (T0) and one month after
  Fatigue measured by Fatigue Severity Scale FSS is a 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree.
  The minimum score is 9 and maximum score possible is 63. Higher is the score, greater is the fatigue severity
Sleep hygiene | Inclusion (T0) and one month after
  Sleep hygiene measured with questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No